CLINICAL TRIAL: NCT06864390
Title: Genicular Nerve Phenol Neurolysis Versus Radiofrequency Ablation for Pain Relief in Grade 4 Knee Osteoarthritis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMASU R17/2025
Record Dates: First submitted 2025-02-14; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Joint Pain
Keywords: phenol neurolysis; radiofrequency; Knee osteoarthritis
MeSH Terms: conditions — Arthralgia; Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- genicular nerve phenol neurolysis (Experimental): chemical neurolysis using 2 mL of 9% phenol solution prepared from crystallized phenol will be applied to each genicular nerve.
  Interventions: Procedure: genicular nerve neurolysis
- genicular nerve radiofrequency ablation (Experimental): Radiofrequency thermocoagulation will be applied to each nerve at 80 degrees for 90 seconds.
  Interventions: Procedure: genicular nerve neurolysis

INTERVENTIONS:
Procedure: genicular nerve neurolysis — The superior medial genicular nerve (SMGN), superior lateral genicular nerve (SLGN), and inferior medial genicular nerve (IMGN) will be blocked either by phenol neurolysis or radiofrequency ablation

SUMMARY:
The goal of this clinical trial is to compare the efficiency and efficacy of genicular nerves blockade by chemical phenol neurolysis versus radiofrequency ablation in managing pain in patients suffering from grade IV KOA in term of NRS pain score.

The participants will be evaluated by numeric rating scale and oxford knee score for assessment of pain relief up to 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Grade 4 knee osteoarthritis according to Kellgren-Lawrence radiological classification.
* Failure to manage pain with conservative methods.

Exclusion Criteria:

* Prior knee replacement
* Patients with cardiac pacemakers or implantable cardiac defibrillators.
* Septic knee or systemic sepsis.
* Allergy to any of the drugs used in the study.
* Coagulopathy or patients on anticoagulants.
* Patients with psychiatric illness.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Numeric rating scale | baseline, 2, 4, 8,12 and 16 weeks after the procedure
  By an independent physician pain will be recorded using numeric rating scale which is a screening tool used to assess pain severity using a 0 - 10 scale with zero meaning no pain and 10 meaning the worst pain ever.

SECONDARY OUTCOMES:
oxford knee score | baseline, 4, 8, 12, 16 weeks after the procedure
  This score is used to assess both function and pain of the knee on a scale ranging from 0 (worst pain and function) and 48 (best function and no pain) this score will be recorded by an independent physician

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Boeith, MD, Principal Investigator — Ain Shams University